CLINICAL TRIAL: NCT04155918
Title: A Phase 2a, Open-Label Study to Evaluate the Safety and Efficacy of AR882 Administered Alone or in Combination With Febuxostat or Allopurinol in Gout Patients
Brief Title: Phase 2a Study of AR882 Alone and in Combination With Febuxostat or Allopurinol in Gout Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arthrosi Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AR882-201
Record Dates: First submitted 2019-10-25; First posted 2019-11-07 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Gout Patients
Keywords: Hyperuricemia; Gout; URAT1
MeSH Terms: conditions — Hyperuricemia; Gout | interventions — Febuxostat; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- AR882/FBX (Experimental)
  Interventions: Drug: Group 1: AR882 Alone and in Combination with Febuxostat (FBX)
- AR882/ALLO (Experimental)
  Interventions: Drug: Group 2: AR882 Alone and in Combination with Allopurinol (ALLO)

INTERVENTIONS:
Drug: Group 1: AR882 Alone and in Combination with Febuxostat (FBX) — AR882 + Febuxostat, AR882 alone, Febuxostat alone
  Other Names: Febuxostat (Adenuric®, Uloric®)
  Arms: AR882/FBX
Drug: Group 2: AR882 Alone and in Combination with Allopurinol (ALLO) — AR882 + Allopurinol, AR882 alone, Allopurinol alone
  Other Names: Allopurinol (Allosig®, Progout®, Zyloprim®)
  Arms: AR882/ALLO

SUMMARY:
The study is designed to evaluate the PK/PD, safety and tolerability of AR882 alone or in combination with febuxostat or allopurinol when administered to gout patients.

ELIGIBILITY:
Key Inclusion Criteria:

* History of gout
* sUA > 7 mg/dL
* Estimated Glomerular Filtration Rate (eGFR) ≥ 60 mL/min/1.73m2

Key Exclusion Criteria:

* Malignancy within 5 years, except for successfully treated basal or squamous cell carcinoma of the skin
* History of cardiac abnormalities
* Active peptic ulcer disease or active liver disease
* History of kidney stones
* Allergy or intolerance to colchicine, febuxostat, and allopurinol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
PD profile of AR882 administered alone or in combination with febuxostat | 22 Days
  Profile from serum uric acid concentration over time
PD profile of AR882 administered alone or in combination with allopurinol | 22 Days
  Profile from serum uric acid concentration over time.
Serum uric acid (sUA) response rate | 22 Days
  sUA response rate to achieve sUA <6, <5, <4, and <3 mg/dL

SECONDARY OUTCOMES:
Area under the curve (AUC) for plasma AR882 | 22 Days
  Profile from plasma in terms of AUC for AR882
Time to maximum plasma concentration (Tmax) for AR882 | 22 Days
  Profile from plasma in terms of Tmax for AR882
Maximum plasma concentration (Cmax) for AR882 | 22 Days
  Profile from plasma in terms of Cmax for AR882
Apparent terminal half-life (t1/2) for AR882 | 22 Days
  Profile from plasma in terms of t1/2 for AR882
Amount excreted (Ae) into urine for AR882 | 22 Days
  Profile from urine in terms of Ae for AR882
Renal clearance (CLr) for AR882 | 22 Days
  Profile from urine in terms of CLr for AR882
AUC for plasma for febuxostat | 22 Days
  Profile from plasma in terms of AUC for febuxostat
Tmax for febuxostat | 22 Days
  Profile from plasma in terms of Tmax for febuxostat
Cmax for febuxostat | 22 Days
  Profile from plasma in terms of Cmax for febuxostat
t1/2 for febuxostat | 22 Days
  Profile from plasma in terms of t1/2 for febuxostat
AUC for plasma allopurinol/oxypurinol | 22 Days
  Profile from plasma in terms of AUC for allopurinol/oxypurinol
Tmax for allopurinol/oxypurinol | 22 Days
  Profile from plasma in terms of Tmax for allopurinol/oxypurinol
Cmax for allopurinol/oxypurinol | 22 Days
  Profile from plasma in terms of Cmax for allopurinol/oxypurinol
t1/2 for for allopurinol/oxypurinol | 22 Days
  Profile from plasma in terms of t1/2 for allopurinol/oxypurinol
Ae in urine for allopurinol/oxypurinol | 22 Days
  Profile from urine in terms of Ae for allopurinol/oxypurinol
CLr for allopurinol/oxypurinol | 22 Days
  Profile from urine in terms of CLr for allopurinol/oxypurinol
AUC for plasma for colchicine | 22 Days
  Profile from plasma in terms of AUC for colchicine
Tmax for colchicine | 22 Days
  Profile from plasma in terms of Tmax for colchicine
Cmax for colchicine | 22 Days
  Profile from plasma in terms of Cmax for colchicine
t1/2 for for colchicine | 22 Days
  Profile from plasma in terms of t1/2 for colchicine
Incidence of Adverse Events, changes in laboratory, electrocardiogram, and vital signs | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Wynne, MBChB, Grad Dip Pharm Med, Principal Investigator — Christchurch Clinical Studies Trust Ltd
Locations (1):
- Christchurch Clinical Studies Trust, Ltd (CCST), Christchurch, New Zealand